CLINICAL TRIAL: NCT01454232
Title: Modification of Human Gut Microbiota in Massive Obesity After Bariatric Surgery: the Role of Energetic Restriction
Brief Title: Adaptation of Human Gut Microbiota to Energetic Restriction
Acronym: microbaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P100111
Record Dates: First submitted 2011-10-07; First posted 2011-10-18 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Obesity; Metabolic Diseases; Nutrition Disorders; Body Weight
Keywords: Obesity; adipose tissue inflammation; Low grade systemic inflammation; gut microbiota; Bariatric surgery
MeSH Terms: conditions — Obesity; Metabolic Diseases; Nutrition Disorders; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- gastric surgery (Other): obese patients addressed for gastric surgery
  Interventions: Other: stools sampling; Other: adipose tissue biopsy
- lean healthy subjects evaluated once (Active Comparator): lean healthy subjects evaluated once
  Interventions: Other: stools sampling; Other: adipose tissue biopsy

INTERVENTIONS:
Other: stools sampling — stools sampling at baseline, 1, 3 and 12 months
Other: adipose tissue biopsy — surgical adipose tissue biopsy during surgery, 1, 3 and 12 months

SUMMARY:
Gut microbiota ecology is altered in obesity and could link obesity and its complications. Bariatric surgery enables a major and sustained weight loss therefore improving obesity related disease.

the investigators primary aim is to evaluate gut microbiota adaptation to weight loss and the specific role of energetic restriction. Furthermore we aim to compare gut flora of obese patients post bariatric surgery to that of lean healthy volunteers.

Thus, the investigators plan to compare gut microbiota from 140 obese individuals before and after either restrictive (gastric banding) procedures or gastric bypass procedures to that of 40 lean healthy volunteers at baseline.

DETAILED DESCRIPTION:
The prevalence of obesity is rising to an epidemic level. Yet medical and pharmacological treatments have proven their limits. Dietetic modifications contribute to adipose tissue alterations and cross talk dysfunction with other tissues linked to weight maintenance. In a previous study in a model of abrupt weight loss 6 months after Roux-en-Y Bypass, the investigators observed a rapid adaptation of the dominant gut microbiota. Conversely some species were directly linked to the improvement of low grade inflammation independently of calory intake.

Therefore the investigators hypothesized that gut microbiota in obese patients could link food consumption with obesity alterations such as metabolic impairments, energetic storage dysfunction and increased systemic and adipose tissue inflammation.

The investigators want to address the specific role of energetic restriction in gut microbiota modification after weight loss.

To answer that question the investigators will evaluate gut microbiota composition before and during the first year after either gastric banding or gastric bypass surgery. they also aim to evaluate whether gut flora post surgery evolves toward that of lean healthy subjects Our study has several objectives. The investigators also aim to assess whether gut microbiota modification is associated with systemic and tissue inflammation reduction and metabolic improvement during the follow up.

This project is based on a clinical protocol performed in massively obese subjects (BMI>40 kg/m²). The investigators plan to recruit 70 obese patients addressed for gastric banding and 70 candidates for gastric bypass. Clinical phenotype, biochemical analysis, body composition, systemic and adipose tissue inflammation, endotoxemia and gut microbiota will be assessed at baseline and 1, 3 and 12 months after surgery. Specific food consumption will be recorded at every time point. A group of 40 lean healthy volunteers will undergo the same phenotyping.

Associations between all these clinical and biological parameters will be assessed at the different point of the follow up.

More generally, this project might lead us to elucidate a new function of gut microbiota and eventually consider novels anti obesity therapeutic strategies

ELIGIBILITY:
Obese group

Inclusion criteria :

* Obesity with BMI> 40 kg/m² or obesity with BMI between 35 and 40 kg/M² with comorbidities (OSA, type 2 diabetes, hypertension etc…)
* Age: 18-65
* women
* weight stable for three months preceding surgery

Exclusion criteria :

* Inflammatory disease
* Pregnancy
* Lactose intolerance
* Antibiotherapy in the three months preceding surgery
* cancer
* Drugs (AINS)

Healthy group

Inclusion criteria :

* 19<BMI<25kg/m²
* Age: 18-65
* women
* non diabetic

Exclusion criteria :

* Inflammatory disease
* Pregnancy
* Antibiotherapy in the two months preceding the visit
* pregnancy
* Drugs (AINS) in the 48h preceding the visit

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-06-07 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Analyse changes early, medium and long term changes in gut microbiota composition in a kinetic manner | at 1, 3 and 12 months after surgery
Compare gut microbiota kinetic changes in obese to gut microbiota healthy volunteers | at 1, 3 and 12 months after surgery in the obese group and compare it to baseline in lean subjects

SECONDARY OUTCOMES:
Establish early, medium and long term changes in insulin sensitivity and GLP1 secretion profile after oral glucose load and look for potential associations between these changes and gut microbiota composition | 1, 3 and 12 months after surgery
Establish early, medium and long term changes in systemic and adipose tissue inflammation and look for potential associations between gut microbiota composition and inflammation modification | 1, 3 and 12 months after surgery
Establish early, medium and long term changes in body composition and look for potential associations between these changes and gut microbiota modifications | 1, 3 and 12 months after surgery
Establish early, medium and long term changes in nutritional blood sample concentrations and look for a potential association between gut microbiota modifications. | 1, 3, 12 months after surgery
Establish early, medium and long term improvement in obesity related disease (reducing the number of treatments and the need for PPC use) and look for potential association with gut microbiota modification | 1, 3 and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Karine Clement, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié Salpêtrière Hospital, Paris, France

REFERENCES:
- [Derived] Torres L, Camila Goncalves Miranda M, Dantas Martins V, Caixeta F, de Almeida Oliveira M, Martins Trindade L, Carvalho de Assis H, Nascimento V, Pinheiro Rosa N, Gomes E, Oliveira Almeida S, Marquet F, Genser L, Marcelin G, Clement K, Russo M, Maria Caetano Faria A, Uceli Maioli T. Obesity-induced hyperglycemia impairs oral tolerance induction and aggravates food allergy. Mucosal Immunol. 2023 Aug;16(4):513-526. doi: 10.1016/j.mucimm.2023.05.008. Epub 2023 Jun 10. PMID 37302712
- [Derived] Aron-Wisnewsky J, Prifti E, Belda E, Ichou F, Kayser BD, Dao MC, Verger EO, Hedjazi L, Bouillot JL, Chevallier JM, Pons N, Le Chatelier E, Levenez F, Ehrlich SD, Dore J, Zucker JD, Clement K. Major microbiota dysbiosis in severe obesity: fate after bariatric surgery. Gut. 2019 Jan;68(1):70-82. doi: 10.1136/gutjnl-2018-316103. Epub 2018 Jun 13. PMID 29899081